CLINICAL TRIAL: NCT07328620
Title: Relationship Between Permissive Hypotension and Acute Kidney Injury in Rhinologic Surgeries: Evaluation With Plasma NGAL and Cystatin C Levels
Brief Title: Is Permissive Hypotension Truly Harmless? Early Biomarker Evidence of Subclinical Kidney Injury in Rhinologic Surgery
Status: Completed | Type: Observational
Sponsor: Gazi University (Other)
Responsible Party: Principal Investigator, Galip Utku Kabacaoglu, M.D., Gazi University
Other Study IDs: PerHypGU0820125
Record Dates: First submitted 2025-12-25; First posted 2026-01-09 (Actual); Last update posted 2026-02-04 (Actual); Status verified 2026-02

CONDITIONS: Acute Kidney Injury; Hypotension
Keywords: Permissive Hypotension; Subclinical Kidney Injury; NGAL; Cystatin C; Rhinologic Surgery; Surgical Field Visibility; Boezaart Score
MeSH Terms: conditions — Acute Kidney Injury; Hypotension

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Days
Biospecimen Retention: Samples Without DNA — Routine perioperative blood samples will be collected, and in addition to standard biochemical tests, NGAL and cystatin C levels will be measured. Cystatin C will be analyzed daily as part of routine clinical workflow, whereas plasma samples for NGAL measurement will be stored at -20°C and analyzed later using a validated ELISA method. No genetic analyses will be performed.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This study aims to investigate the effects of permissive hypotension, which is routinely used in rhinologic surgeries such as rhinoplasty, septoplasty, and functional endoscopic sinus surgery (FESS), on renal function. Although permissive hypotension has been widely practiced to improve surgical field visibility and reduce intraoperative blood loss, its specific definition is not standardized in the literature. In most studies, maintaining mean arterial pressure (MAP) within the range of 50-65 mmHg is considered permissive hypotension. MAP values below 60 mmHg have been associated with increased risk of cardiac and renal complications. However, in otherwise healthy patients, such episodes are frequently tolerated without clinically apparent renal dysfunction.

The kidneys have a strong compensatory reserve capacity, and early tubular injury may not be detected by conventional renal function tests such as serum creatinine. Therefore, the use of more sensitive biomarkers is necessary to detect potential subclinical injury.

In this prospective observational study, plasma NGAL and cystatin C levels will be measured from routine preoperative and postoperative (12-24 hours) blood samples obtained from adult patients undergoing rhinologic procedures. A ≥25% increase in these biomarkers from baseline will be considered indicative of subclinical acute kidney injury.

Additionally, intraoperative hemodynamic data will be monitored, and the duration of MAP <60 mmHg and MAP <65 mmHg will be recorded. At the end of the procedure, surgical field conditions will be evaluated using the Boezaart Surgical Field Score. The relationship between these parameters and biomarker changes will be analyzed.

The goal of this study is to determine whether early, clinically silent renal injury may occur during permissive hypotension and to provide insight into its potential implications for future renal function. All interventions and blood samplings are part of routine care, and no additional procedures will be performed for research purposes.

DETAILED DESCRIPTION:
Permissive hypotension is a commonly used anesthetic technique in rhinologic surgeries to optimize surgical conditions by reducing bleeding and improving visualization. Although widely applied, a standardized definition is lacking in the literature. Many studies define permissive hypotension as maintaining mean arterial pressure (MAP) between 50-65 mmHg. MAP values lower than 60 mmHg may compromise tissue perfusion and oxygenation, particularly in the renal medulla, possibly predisposing patients to ischemic stress. Despite this, in patients without significant comorbidities, these controlled reductions typically do not result in clinically evident kidney dysfunction, which supports the continued use of this technique in suitable cases.

However, due to the high renal reserve, subclinical kidney injury may still occur without notable changes in serum creatinine or urine output. The early detection of renal injury may be possible through biomarkers such as neutrophil gelatinase-associated lipocalin (NGAL) and cystatin C, which are more sensitive to structural renal injury. This study is designed to evaluate such potential biomarker changes during permissive hypotension applied for rhinologic surgery.

Study Design and Methods: This is a prospective observational, single-center study including 35 adult patients aged 18-65 years who are scheduled to undergo elective rhinoplasty, septoplasty, or FESS. Patients with a history of chronic kidney disease, uncontrolled hypertension or diabetes mellitus, or contraindications to hypotensive anesthesia will be excluded. Informed consent will be obtained preoperatively. All blood sampling and hemodynamic monitoring will be performed as part of routine clinical care, and no additional intervention will be introduced.

Data Collection and Measurements: Preoperative routine blood samples will be analyzed for renal biomarkers including plasma NGAL and cystatin C, in addition to standard biochemistry profiles. Plasma NGAL levels will be measured using a validated ELISA method (Elabscience, USA), and plasma cystatin C levels will be analyzed using a particle-enhanced turbidimetric assay (Siemens Atellica Neph 630).

Intraoperative hemodynamic variables will be recorded every 5 minutes throughout anesthesia, and total durations of MAP <60 mmHg and MAP <65 mmHg will be calculated. Postoperatively, between 12 and 24 hours, routine blood sampling will again be performed, and NGAL and cystatin C levels will be re-evaluated. At the end of surgery, surgical field visibility will be assessed by the otorhinolaryngology surgical team using the Boezaart Surgical Field Score.

Outcome Measures: The primary outcome of this study is the presence of subclinical renal injury, defined as a ≥25% increase in plasma NGAL and/or cystatin C from preoperative baseline to the postoperative 12-24-hour measurement. Secondary outcomes include the association between biomarker changes and intraoperative hypotension exposure (duration of MAP <60 mmHg and MAP <65 mmHg), as well as the relationship between hypotension and surgical field quality assessed with the Boezaart Score.

Safety and Adverse Event Monitoring: All procedures are routine clinical practices and carry no additional risk to participants. In the event of postoperative impairment of renal function, standard clinical management will be followed, including fluid optimization and nephrology consultation when appropriate.

Data Confidentiality: All collected data will be de-identified and stored securely with restricted access limited to the research team.

ELIGIBILITY:
Inclusion Criteria:

* Adults aged 18-65 years
* Scheduled for elective rhinologic surgery (rhinoplasty, septoplasty, or functional endoscopic sinus surgery)
* ASA physical status I-II
* Able to provide written informed consent
* Undergoing controlled hypotension anesthesia as part of routine clinical management

Exclusion Criteria:

* Known chronic kidney disease (baseline creatinine above normal range or documented CKD)
* Uncontrolled hypertension or uncontrolled diabetes mellitus
* Contraindications to controlled hypotensive anesthesia
* Pregnant or breastfeeding women
* History of major cardiovascular disease affecting renal perfusion (e.g., severe heart failure)
* Use of nephrotoxic medications preoperatively that may interfere with renal biomarker interpretation
* Perioperative complications requiring deviation from routine anesthetic management (e.g., major bleeding or hemodynamic instability)

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Adult patients aged 18-65 years undergoing elective rhinologic surgery under controlled hypotension anesthesia at a single tertiary care center will be enrolled. The study population consists of otherwise healthy individuals (ASA I-II) without known kidney disease and without major comorbidities that could independently affect renal function.
Sampling Method: Non-Probability Sample
Enrollment: 35 (Actual)
Dates: Start 2025-03-01 (Actual); Primary Completion 2025-05-30 (Actual); Study Completion 2025-07-30 (Actual)

PRIMARY OUTCOMES:
Change in plasma NGAL and cystatin C concentrations indicating subclinical kidney injury | Preoperative baseline to postoperative 12-24 hours
  Plasma neutrophil gelatinase-associated lipocalin (NGAL) concentration (ng/mL) measured by ELISA assay and plasma cystatin C concentration (mg/L) measured by automated nephelometric assay will be assessed preoperatively and at postoperative 12-24 hours.
  A relative increase of ≥25% from baseline in either biomarker will be used to define subclinical renal injury.

SECONDARY OUTCOMES:
Duration of mean arterial pressure below 60 mmHg during anesthesia | Intraoperative period
  The total duration (minutes) of intraoperative mean arterial pressure (MAP) <60 mmHg recorded at 5-minute intervals from standard anesthesia monitoring.
Duration of mean arterial pressure below 65 mmHg during anesthesia | Intraoperative period
  The total duration (minutes) of intraoperative mean arterial pressure (MAP) <65 mmHg recorded at 5-minute intervals from standard anesthesia monitoring.
Correlation between intraoperative hypotension duration and renal biomarker changes | Intraoperative period to postoperative 12-24 hours
  Correlation between cumulative duration of MAP <60 mmHg and <65 mmHg (minutes) and percentage change in plasma NGAL (ng/mL) and cystatin C (mg/L) concentrations from baseline.
Correlation between surgical field quality and intraoperative hypotension | End of surgery
  Correlation between Boezaart Surgical Field Score (0-5 scale) and cumulative duration of MAP <60 mmHg and <65 mmHg (minutes).

CONTACTS AND LOCATIONS:
Overall Officials: Hasan K Pampal, M.D., Study Director — Gazi University Faculty of Medicine, Department of Anesthesiology and Reanimation
Locations (1):
- Gazi University Faculty of Medicine, Ankara, Yenimahalle, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
Individual participant data (IPD) will not be shared. Only de-identified, aggregated study results will be made available through scientific publications and presentations.

REFERENCES:
- [Background] Salmasi V, Maheshwari K, Yang D, Mascha EJ, Singh A, Sessler DI, Kurz A. Relationship between Intraoperative Hypotension, Defined by Either Reduction from Baseline or Absolute Thresholds, and Acute Kidney and Myocardial Injury after Noncardiac Surgery: A Retrospective Cohort Analysis. Anesthesiology. 2017 Jan;126(1):47-65. doi: 10.1097/ALN.0000000000001432. PMID 27792044
- [Background] Petrova I, Alexandrov A, Vladimirov G, Mateev H, Bogov I, Paskaleva I, Gotcheva N. NGAL as Biomarker of Clinical and Subclinical Damage of Kidney Function after Coronary Angiography. Diagnostics (Basel). 2023 Mar 20;13(6):1180. doi: 10.3390/diagnostics13061180. PMID 36980488
- [Background] Sessler DI, Bloomstone JA, Aronson S, Berry C, Gan TJ, Kellum JA, Plumb J, Mythen MG, Grocott MPW, Edwards MR, Miller TE; Perioperative Quality Initiative-3 workgroup; POQI chairs; Miller TE, Mythen MG, Grocott MP, Edwards MR; Physiology group; Preoperative blood pressure group; Intraoperative blood pressure group; Postoperative blood pressure group. Perioperative Quality Initiative consensus statement on intraoperative blood pressure, risk and outcomes for elective surgery. Br J Anaesth. 2019 May;122(5):563-574. doi: 10.1016/j.bja.2019.01.013. Epub 2019 Feb 27. PMID 30916004
- [Background] Ostermann M, Legrand M, Meersch M, Srisawat N, Zarbock A, Kellum JA. Biomarkers in acute kidney injury. Ann Intensive Care. 2024 Sep 15;14(1):145. doi: 10.1186/s13613-024-01360-9. PMID 39279017
- [Background] Khetpal S, Elias A, Alford J, et al. Anesthesia for rhinoplasty: a summary of clinical considerations, therapeutic modalities, outcomes, and future directions. JCA Adv. 2024;1:100040. doi:10.1016/j.jcadva.2024.100040.